CLINICAL TRIAL: NCT00781872
Title: Explorative Trial to Investigate the Safety and Clinical Effects of Autologous Mesenchymal Bone Marrow Stem Cells (MSC) Following Their Intrathecal and Intravenous Administration in Severe Cases of Multiple Sclerosis (MS)
Brief Title: Mesenchymal Stem Cells for the Treatment of MS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Dimitrios Karussis, Head of The Center for Multiple Sclerosis & Unit of Neuroimmunology, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS22MSC-HMO-CTIL
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis (MS); bone marrow stromal cells; stem cells
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with autologous mesenchymal stem cells (MSC) intrathecally and intravenously (Experimental): Intrathecal and intravenous treatment with autologous mesenchymal stem cells (MSC) intrathecally and intravenously in patients with active multiple sclerosis, failures to respond to other treatments
  Interventions: Biological: Injection of autologous bone marrow derived mesenchymal stem cells

INTERVENTIONS:
Biological: Injection of autologous bone marrow derived mesenchymal stem cells — 60 million cells intrathecally (approximately 1 million cells per Kg of body weight) and 20 million cells intravenously
  Other Names: Mesenchymal stem cells of bone marrow

SUMMARY:
Although, effective immunotherapies for MS exist which downregulate the anti-myelin reactivity and reduce the rate of relapses of the disease, there is no effective means today to stop the progression of disability and induce remyelination. Neuronal stem cells were shown to possess the ability to restore neuronal activity and produce new neurons through transdifferentiation. Various other types of stem cells were tested in animal models with promising results, revealing a potential for restoration of the neurological function in neuroimmune and neurodegenerative conditions. Adult bone marrow derived stromal cells (MSC) were shown to induce similar (to neuronal stem cells) immunomodulatory and neuroregenerative effects and were shown in our laboratory to induce neuroprotection in the animal model of chronic experimental autoimmune encephalomyelitis (EAE). MSCs offer practical advantages for clinical therapeutic applications, since they can be obtained from the adult bone marrow and therefore the patient can be the donor for himself, without any danger for rejection of the cells. In addition, MSCs carry a safer profile and are less prone to malignant transformation.

Our initial clinical experience with 10 patients with ALS and 10 with multiple sclerosis show that intravenous and intrathecal administration of MSCs is feasible and safe.

In this study we propose an explorative protocol with the injection of MSCs (both intrathecally and intravenously) in patients with MS, in an effort to prevent further neurodegeneration through neuroprotective mechanisms and induce neuroregeneration and restoration of neuronal function.

The primary endpoint will be to further evaluate the safety and feasibility of the treatment with MSC infusions, in MS patients. Additionally, the migration ability of the transplanted cells will be evaluated by tagging MSCs with the superparamagnetic iron oxide particle (Feridex) for detection by MRI. Clinically the patients will be followed by monthly evaluations of the MS functional rating scale (EDSS) scale. The MRI, will be also used to evaluate changes in the total volume of lesions in the brain and the degree of atrophy.

Significance: This project may provide information for possible therapeutic uses of this type of bone marrow adult stem cells in MS but may also serve as a pilot platform and pave the path for future applications of various types of stem cells in neurodegerative diseases, in general.

DETAILED DESCRIPTION:
This study, is designed as a phase 1/2 open-safety clinical trial. At its first phase, 15 consenting patients with MS are included.

Inclusion Criteria:

Consenting patients fulfilled the following 4 inclusion criteria for this study:

1. the clinical criteria of Poser et alfor definite MS;
2. men and nonpregnant women aged 25 to 65 years;
3. duration of disease longer than 5 years; and
4. failure to respond to the currently available and registered agents for MS (ie, interferons, glatiramer acetate [Copaxone], and immuno-suppressors), as manifested by an increase of at least 1 degree in the EDSS score during the past year or the appearance of at least 2 major MS relapses during the same period.

Exclusion criteria:

1. patients who were treated with cytotoxic medications (ie, cyclophosphamide, mitoxantrone, and azathioprine) during the 3 months before the trial;
2. patients with significant cardiac, renal, or hepatic failure or any other disease that may interfere with the ability to interpret the results of the study;
3. patients with an active infection; and
4. patients who showed severe cognitive decline or were unable to understand and sign the informed consent.

Bone marrow aspiration is performed under short general anesthesia with puncture from the posterior superior iliac crest while the patient was lying in a left or a right lateral position. Approximately 200 mL of bone marrow inocula are obtained from each patient.

MSC Preparation and Culture A culture of purified MSCs is prepared under aseptic conditions (positively pressurized clean rooms) using filtered sterilized Dulbecco modified Eagle medium with low glucose lev- els (Qiagen, Valencia, California) supplemented with 10% fetal bovine serum, 1% L-glutamine, and 1% penicillin-streptomycin- nystatin solution (all from Biological Industries, Kibbutz Beit- Haemek, Israel).

Mesenchymal cells are cultured for 40 to 60 days, until they reach confluency, and then harvested and cryopreserved in 10% dimethyl sulfoxide-containing medium in liquid nitrogen (-196°C). At 2 weeks, a sample is taken for sterility testing and quality control. After sterility confirmed, the MSCs are transferred to the laboratory on dry ice, thawed in a 37°C water bath, and washed twice with normal saline solution to remove any residual dimethyl sulfoxide. The cells are then resuspended in normal saline at a concentration of 10x106/mL to 15x106/mL. Two-thirds of the total number of cells (usually 60x106 to 100x106) are injected intrathecally, and one-third, intravenously. A sample of the cells to be injected is tested by fluorescence-activated cell sorter (FACS) analysis; cells (98%) should express the surface markers characteristic of MSCs (CD29, CD73, CD90, CD105, and CD166) and be negative for CD34, CD45, and CD14.

Treatment Protocol All patients receive an intrathecal injection via a standard lumbar puncture (mean of 1 million cells per Kg of body weight) and an intravenous injection of 0.3-1 million cells per kg, intravenously..

An extension phase is scheduled for patients completing the first phase of this trial as an open prospective study with repeated intrathecal or intravenous injections of autologous MSC in patients from the initial trial and 10 additional ones (total up to 24 patients) with progressive forms of MS (secondary progressive, primary progressive or relapsing-progressive). Patients should be defined as failures to first and second lines of immunomodulatory treatments experiencing deterioration (at least 0.5 degree in the EDSS scale) during the year preceding their inclusion to our study or had at least one major relapse without sufficient recovery. Patients will be treated with 1x10 million MSC per kg of body weight, intrathecally and intravenously and subsequently with up to 8 courses of IT- or IV-injections of MSC (at the same dose), at intervals of 6-12 months. The duration of the trial is 4 years.

Patients will be followed up every 3 months for the whole duration of the trial, for safety assessment and changes in the disability scores (EDSS).

Immunological analysis will be performed at 4 time points (day 1, month 1, month 3 and month 6) following the first MSC-treatment and will include a fluorescent cell sorter (FACS) analysis to evaluate the proportions of the lymphocytes expressing markers of immune activation or of regulatory cell phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting patients fulfilling the Poser's clinical criteria for definite MS
2. Age: 35-65, males and females
3. Duration of disease: >5 years
4. Failure to the currently available -registered- for MS immunomodulatory treatments (ie interferons, Copaxone, immunosuppression): the lack of response to (at least two) of these treatments will be determined/defined by either an increase (deterioration) of at least one degree in the EDSS score during the last year or the appearance of at least two major relapses of MS during the same period of time (under treatment).

Exclusion criteria

1. Patients who were treated with cytotoxic medications (cyclophosphamide, Mitoxanthrobne etc) during the last 3 months prior to the inclusion
2. Patients suffering from significant cardiac, renal or hepatic failure or any other disease that may risk the patient or interfere with the ability to interpret the results
3. Patients with active infections
4. Patients with severe cognitive decline or inability to understand and sign the informed consent

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety of one or multiple intrathecaland intravenous injections of autologous MSC in Multiple sclerosis | One year for the first phase; 4 years for the extension phase
  Appearance of adverse events during the 1-4 years of follow up after one or multiple treatments with MSC

SECONDARY OUTCOMES:
Clinical effects in terms of changes in the expended disability status scale (EDSS) at 3-6 month intervals | One year for the first phase; 4 years for the extension phase
  The changes in EDSS score and relapses will be recorded at 3-6 month intervals in patients treated with 1-8 treatments of MSC interthecally and intravenously
Immunological effects of treatment with MSC in MS | 1-6 months after the first treatment with MSC
  Changes in the proportion of T-regs (CD4/CD25/FoxP3) and of activated cells (CD69) and the proliferation ability of lymphocytes in patients' peripheral blood at 1 day, 1, 3 and 6 months following the first treatment with MSC (compared to baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karussis, Prof., Principal Investigator — Hadassah Medical Organization

REFERENCES:
- [Derived] Karussis D, Karageorgiou C, Vaknin-Dembinsky A, Gowda-Kurkalli B, Gomori JM, Kassis I, Bulte JW, Petrou P, Ben-Hur T, Abramsky O, Slavin S. Safety and immunological effects of mesenchymal stem cell transplantation in patients with multiple sclerosis and amyotrophic lateral sclerosis. Arch Neurol. 2010 Oct;67(10):1187-94. doi: 10.1001/archneurol.2010.248. PMID 20937945